CLINICAL TRIAL: NCT01662999
Title: A Single-dose, Open-label, Randomized, 3 Period, 3 Treatment Crossover Study to Evaluate the Pharmacokinetics of Saxagliptin 5 mg and Dapagliflozin 10 mg When Coadministered to Fasted Healthy Subjects
Brief Title: Drug Interaction Study of Saxagliptin in Combination With Dapagliflozin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CV181-191
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Results first posted 2013-12-23 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- A-B-C: Saxagliptin-Dapagliflozin-(Saxagliptin+Dapagliflozin) (Experimental): Treatment A: Saxagliptin 5mg, Tablet, Oral; Single dose Treatment B: Dapagliflozin 10mg, Tablet, Oral; single dose Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral; single dose
  Interventions: Drug: Saxagliptin; Drug: Dapagliflozin
- A-C-B: Saxagliptin-(Saxagliptin+Dapagliflozin)-Dapagliflozin (Experimental): Treatment A: Saxagliptin 5mg, Tablet, Oral, single dose; Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral, single dose; Treatment B: Dapagliflozin 10mg, Tablet, Oral, single dose
  Interventions: Drug: Saxagliptin; Drug: Dapagliflozin
- B-A-C: Dapagliflozin-Saxagliptin-(Saxagliptin+Dapagliflozin) (Experimental): Treatment B: Dapagliflozin 10mg, Tablet, Oral, single dose. Treatment A: Saxagliptin 5mg, Tablet, Oral, single dose; Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral, single dose
  Interventions: Drug: Saxagliptin; Drug: Dapagliflozin
- B-C-A: Dapagliflozin-(Saxagliptin+Dapagliflozin)-Saxagliptin (Experimental): Treatment B: Dapagliflozin 10mg, Tablet, Oral, single dose; Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral, single dose; Treatment A: Saxagliptin 5mg, Tablet, Oral, single dose
  Interventions: Drug: Saxagliptin; Drug: Dapagliflozin
- C-A-B: (Saxagliptin+Dapagliflozin)-Saxagliptin-Dapagliflozin (Experimental): Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral, single dose; Treatment A: Saxagliptin 5mg, Tablet, Oral, single dose; Treatment B: Dapagliflozin 10mg, Tablet, Oral, single dose
  Interventions: Drug: Saxagliptin; Drug: Dapagliflozin
- C-B-A: (Saxagliptin+Dapagliflozin)-Dapagliflozin-Saxagliptin (Experimental): Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral, single dose; Treatment B: Dapagliflozin 10mg, Tablet, Oral, Once daily, single dose; Treatment A: Saxagliptin 5mg, Tablet, Oral, single dose
  Interventions: Drug: Saxagliptin; Drug: Dapagliflozin

INTERVENTIONS:
Drug: Saxagliptin
  Other Names: Onglyza®; BMS-477118
Drug: Dapagliflozin
  Other Names: BMS-512148

SUMMARY:
The purpose of this study is to evaluate whether the pharmacokinetics (body concentrations/metabolism of the drug) of Saxagliptin and Dapagliflozin are affected when they are administered together

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by no clinically significant deviation from normal in medical history, Physical Examination, vital signs, 12-lead ECG, and clinical laboratory determinations
* Body mass index (BMI) of 18 to 30 kg/m2
* Men and women, ages 18 to 45 years
* Women of childbearing potential must use acceptable methods of highly effective birth control

Exclusion Criteria:

* History of chronic or recurrent urinary tract infection for females
* History of allergies or adverse reactions to Dipeptidyl peptidase-IV (DPP4) or Sodium-glucose transporter type 2 (SGLT2) inhibitors
* Any significant acute or chronic medical illness
* Current or recent gastrointestinal disease
* Any major surgery within 4 weeks of study drug administration
* Prior exposure to saxagliptin or dapagliflozin or related drugs

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Icon Clinical Pharmacology, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Vakkalagadda B, Lubin S, Reynolds L, Liang D, Marion AS, LaCreta F, Boulton DW. Lack of a Pharmacokinetic Interaction Between Saxagliptin and Dapagliflozin in Healthy Subjects: A Randomized Crossover Study. Clin Ther. 2016 Aug;38(8):1890-9. doi: 10.1016/j.clinthera.2016.07.005. Epub 2016 Aug 2. PMID 27491280
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 August 2012 to 29 November 2012. Phase 1 Clinical Pharmacology center with healthy, fasted participants.
Pre-assignment Details: 89 participants enrolled; 42 randomized and treated with study drug. 47 not randomized for following reasons: 3 withdrew consent, 38 no longer met study criteria, 6 had other reasons. Treatment was administered on Day 1 of each period after fast of 10 hours; Washout began after single dose in the period and was for at least 6 days.
Groups:
- A-B-C: Saxagliptin-Dapagliflozin-(Saxagliptin+Dapagliflozin): Single dose of:
  Treatment A: Saxagliptin 5mg, Tablet, Oral; Treatment B: Dapagliflozin 10mg, Tablet, Oral; Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral
- A-C-B: Saxagliptin-(Saxagliptin+Dapagliflozin)-Dapagliflozin: Single dose of:
  Treatment A: Saxagliptin 5mg, Tablet, Oral; Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral; Treatment B: Dapagliflozin 10mg, Tablet, Oral
- B-A-C: Dapagliflozin-Saxagliptin-(Saxagliptin+Dapagliflozin): Single dose of:
  Treatment B: Dapagliflozin 10mg, Tablet, Oral; Treatment A: Saxagliptin 5mg, Tablet, Oral; Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral
- B-C-A: Dapagliflozin-(Saxagliptin+Dapagliflozin)-Saxagliptin: Single dose of:
  Treatment B: Dapagliflozin 10mg, Tablet, Oral; Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral; Treatment A: Saxagliptin 5mg, Tablet, Oral
- C-A-B: (Saxagliptin+Dapagliflozin)-Saxagliptin-Dapagliflozin: Single dose of:
  Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral; Treatment A: Saxagliptin 5mg, Tablet, Oral; Treatment B: Dapagliflozin 10mg, Tablet, Oral
- C-B-A: (Saxagliptin+Dapagliflozin)-Dapagliflozin-Saxagliptin: Single dose of:
  Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral; Treatment B: Dapagliflozin 10mg, Tablet, Oral; Treatment A: Saxagliptin 5mg, Tablet
Period: Period 1
Arm/Group | A-B-C: Saxagliptin-Dapagliflozin-(Saxagliptin+Dapagliflozin) | A-C-B: Saxagliptin-(Saxagliptin+Dapagliflozin)-Dapagliflozin | B-A-C: Dapagliflozin-Saxagliptin-(Saxagliptin+Dapagliflozin) | B-C-A: Dapagliflozin-(Saxagliptin+Dapagliflozin)-Saxagliptin | C-A-B: (Saxagliptin+Dapagliflozin)-Saxagliptin-Dapagliflozin | C-B-A: (Saxagliptin+Dapagliflozin)-Dapagliflozin-Saxagliptin
Started | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | A-B-C: Saxagliptin-Dapagliflozin-(Saxagliptin+Dapagliflozin) | A-C-B: Saxagliptin-(Saxagliptin+Dapagliflozin)-Dapagliflozin | B-A-C: Dapagliflozin-Saxagliptin-(Saxagliptin+Dapagliflozin) | B-C-A: Dapagliflozin-(Saxagliptin+Dapagliflozin)-Saxagliptin | C-A-B: (Saxagliptin+Dapagliflozin)-Saxagliptin-Dapagliflozin | C-B-A: (Saxagliptin+Dapagliflozin)-Dapagliflozin-Saxagliptin
Started | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 7 | 7 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | A-B-C: Saxagliptin-Dapagliflozin-(Saxagliptin+Dapagliflozin) | A-C-B: Saxagliptin-(Saxagliptin+Dapagliflozin)-Dapagliflozin | B-A-C: Dapagliflozin-Saxagliptin-(Saxagliptin+Dapagliflozin) | B-C-A: Dapagliflozin-(Saxagliptin+Dapagliflozin)-Saxagliptin | C-A-B: (Saxagliptin+Dapagliflozin)-Saxagliptin-Dapagliflozin | C-B-A: (Saxagliptin+Dapagliflozin)-Dapagliflozin-Saxagliptin
Started | 7 | 7 | 7 | 7 | 7 | 7
Completed | 7 | 6 (Participant did not provide 36, 48, or 60 hour samples in this period for Treatment B.) | 7 | 7 | 7 | 7
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- A-B-C: Saxagliptin-Dapagliflozin-(Saxagliptin+Dapagliflozin): Treatment A: Saxagliptin 5mg, Tablet, Oral; Treatment B: Dapagliflozin 10mg, Tablet, Oral; Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral.
- A-C-B: Saxagliptin-(Saxagliptin+Dapagliflozin)-Dapagliflozin: Treatment A: Saxagliptin 5mg, Tablet, Oral; Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral; Treatment B: Dapagliflozin 10mg, Tablet, Oral.
- B-A-C: Dapagliflozin-Saxagliptin-(Saxagliptin+Dapagliflozin): Treatment B: Dapagliflozin 10mg, Tablet, Oral; Treatment A: Saxagliptin 5mg, Tablet, Oral; Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral
- B-C-A: Dapagliflozin-(Saxagliptin+Dapagliflozin)-Saxagliptin: Treatment B: Dapagliflozin 10mg, Tablet, Oral; Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral; Treatment A: Saxagliptin 5mg, Tablet, Oral.
- C-A-B: (Saxagliptin+Dapagliflozin)-Saxagliptin-Dapagliflozin: Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets,Oral; Treatment A: Saxagliptin 5mg, Tablet, Oral; Treatment B: Dapagliflozin 10mg, Tablet, Oral.
- C-B-A: (Saxagliptin+Dapagliflozin)-Dapagliflozin-Saxagliptin: Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral; Treatment B: Dapagliflozin 10mg, Tablet, Oral; Treatment A: Saxagliptin 5mg, Tablet, Oral.
- Total: Total of all reporting groups
Arm/Group | A-B-C: Saxagliptin-Dapagliflozin-(Saxagliptin+Dapagliflozin) | A-C-B: Saxagliptin-(Saxagliptin+Dapagliflozin)-Dapagliflozin | B-A-C: Dapagliflozin-Saxagliptin-(Saxagliptin+Dapagliflozin) | B-C-A: Dapagliflozin-(Saxagliptin+Dapagliflozin)-Saxagliptin | C-A-B: (Saxagliptin+Dapagliflozin)-Saxagliptin-Dapagliflozin | C-B-A: (Saxagliptin+Dapagliflozin)-Dapagliflozin-Saxagliptin | Total
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 7 | 7 | 7 | 7 | 42
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (6.47) | 28.7 (5.02) | 27.7 (6.99) | 32.0 (6.51) | 34.4 (5.74) | 33.3 (7.95) | 32.0 (6.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 3 | 2 | 2 | 13
  Male | 5 | 5 | 5 | 4 | 5 | 5 | 29
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 7 | 7 | 7 | 7 | 42
Body Surface Area (m^2) [Mean (Standard Deviation); unit: m^2] — Body surface area was measured in meters squared (m^2) prior to first dose of study drug (Day -1).
  m^2 | 1.90 (0.187) | 1.92 (0.145) | 1.91 (0.208) | 1.95 (0.170) | 1.94 (0.166) | 1.85 (0.108) | 1.91 (0.160)
Body Weight (kg) [Mean (Standard Deviation); unit: kg] — Body weight was measured in kilograms (k) prior to first dose of study drug (Day -1).
  kg | 77.94 (12.250) | 78.94 (8.100) | 76.01 (14.589) | 80.73 (11.903) | 79.64 (11.223) | 71.71 (6.404) | 77.50 (10.813)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Dapagliflozin From a Single Dose of Dapagliflozin Versus Cmax of Dapagliflozin From Co-administered Saxagliptin Plus Dapagliflozin - Pharmacokinetic Evaluable Population
Description: The geometric mean of the maximum observed plasma concentration (Cmax) is presented below; serial blood samples for determination of study drug were collected predose (0 hours (h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h,and 60 h postdose, relative to dosing on Day 1 in each cross over period and these data are summarized in the Pharmacokinetic (PK) parameter of Cmax presented here. Plasma samples were analyzed for dapagliflozin by High Performance Liquid chromatography-Mass Spectrometry (HPLC-MS/MS) using a validated method; nominal range of 0.200 to 100 nanograms per milliliter (ng/mL). Dapagliflozin Cmax was derived from plasma concentration versus time data using a non-compartmental method, using a validated PK analysis program ™. Actual sampling times were used for PK calculations. Cmax was reported in ng/mL.
Time Frame: Day 1 (0 h to 60 h post dose) in each period
Population: Pharmacokinetic (PK) Evaluable: All participants who received at least 1 dose of any study drug and had at least 1 valid PK parameter for at least 1 analyte. One participant in the ACB treatment sequence withdrew consent after having received all 3 treatments; this participant did not provide 36-, 48-, or 60-hour samples in Period 3 (Treatment B).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 10 mg Dapagliflozin: Treatment B: Single dose oral tablet of 10 mg Dapagliflozin
- 5 mg Saxagliptin + 10 mg Dapagliflozin: Treatment C: Co-administration of a single dose oral tablet of 10 mg Dapagliflozin plus a single dose of oral tablet of 5mg saxagliptin.
Arm/Group | 10 mg Dapagliflozin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 41 | 42
ng/mL | 133 (23) | 125 (27)
Statistical Analysis 1: Comparison: 10 mg Dapagliflozin vs 5 mg Saxagliptin + 10 mg Dapagliflozin; The statistical model includes treatment and period as fixed effects and measurements within each participant as repeated measurements. The adjusted geometric means are from the mixed model; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric mean = 0.943, 90% CI 2-sided [0.867 to 1.026]

2. Primary Outcome: Area Under the Concentration-time Curve (AUC) From Time Zero to Infinity [AUC(INF)] of Dapagliflozin From a Single Dose of Dapagliflozin Versus AUC (INF) of Dapagliflozin When Co-administered With Saxagliptin - PK Evaluable Population
Description: AUC(INF) is area under the plasma concentration-time curve from time 0 extrapolated to infinity. Serial blood samples for determination of study drug were collected predose (0 hours (h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Plasma samples were analyzed for dapagliflozin by HPLC-MS/MS using a validated method; nominal range of 0.200 to 100 nanograms per milliliter (ng/mL). Actual sampling times were used for PK calculations. AUC(INF) was derived from the plasma concentration versus time profile for study drug using a validated PK analysis program ™ and was measured in nanograms*hours per milliliter (ng*h/mL).
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: PK Evaluable Population: All participants who received at least 1 dose of any study drug and had at least 1 valid PK parameter for at least 1 analyte. One participant in the ACB treatment sequence withdrew consent after having received all 3 treatments; this participant did not provide 36-, 48-, or 60-hour samples in Period 3 (Treatment B).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 10 mg Dapagliflozin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 41 | 42
ng*h/mL | 547 (23) | 539 (20)
Statistical Analysis 1: Comparison: 10 mg Dapagliflozin vs 5 mg Saxagliptin + 10 mg Dapagliflozin; Treatment B versus C in AUC(INF). The statistical model includes treatment and period as fixed effects and measurements within each participant as repeated measurements. The adjusted geometric means are from the mixed model; Test type: Superiority or Other; Mixed Models Analysis; Ration of adjusted geometric mean = 0.984, 90% CI 2-sided [0.961 to 1.008]

3. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of Dapagliflozin From a Single Dose of 10 mg Dapagliflozin Versus Tmax of Dapagliflozin When Co-administered With 5 mg Saxagliptin - PK Evaluable Population
Description: Serial blood samples for determination of study drug were collected predose (0 h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Plasma samples were analyzed for dapagliflozin by HPLC-MS/MS using a validated method. Actual sampling times were used for PK calculations. Tmax was derived from the plasma concentration versus time profile using a validated PK analysis program ™ and was measured in hours.
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: PK Evaluable Population: All participants who received at least 1 dose of any study drug and had at least 1 valid PK parameter for at least 1 analyte. 1 participant (ACB treatment sequence) withdrew consent after having received all 3 treatments and did not provide 36-, 48-, or 60-hour samples in Period 3 (Treatment B). This did not impact T-HALF.
Measure: Median (Full Range); unit: hours
Arm/Group | 10 mg Dapagliflozin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 41 | 42
hours | 1.00 [0.50 to 2.02] | 1.00 [0.50 to 2.00]

4. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration AUC(0-T) of Dapagliflozin From a Single Dose of 10 mg Dapagliflozin Versus AUC(0-T) for Dapagliflozin When Co-administered With 5 mg Saxagliptin
Description: AUC(0-T) is area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (linear up/log down trapezoidal method). Serial blood samples for determination of study drug were collected predose (0 h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Plasma samples were analyzed for dapagliflozin by HPLC-MS/MS using a validated method; nominal range of 0.200 to 100 nanograms per milliliter (ng/mL). Actual sampling times were used for PK calculations. AUC(0-T) was derived from the plasma concentration versus time profile for study drug using a validated PK analysis program ™ and was measured in nanograms*hours per milliliter (ng*h/mL).
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 10 mg Dapagliflozin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 41 | 42
ng*h/mL | 529 (23) | 523 (19)
Statistical Analysis 1: Comparison: 10 mg Dapagliflozin vs 5 mg Saxagliptin + 10 mg Dapagliflozin; Treatment B versus C in AUC(0-T). The statistical model includes treatment and period as fixed effects and measurements within each participant as repeated measurements. The adjusted geometric means are from the mixed model; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric mean = 0.990, 90% CI 2-sided [0.966 to 1.014]

5. Secondary Outcome: Half-life (T-HALF) of Dapagliflozin From a Single Dose of Dapagliflozin Versus T-Half of Dapagliflozin When Co-administered With Saxagliptin - PK Evaluable Population
Description: Serial blood samples for determination of study drug were collected predose (0 h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Plasma samples were analyzed for dapagliflozin by HPLC-MS/MS using a validated method. Actual sampling times were used for PK calculations. T-HALF was derived from the plasma concentration versus time profile using a validated PK analysis program ™ and was measured in hours.
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Groups:
- 10mg Dapagliflozin: Treatment B: Single dose oral tablet of 10 mg Dapagliflozin
Arm/Group | 10mg Dapagliflozin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 42 | 42
hours | 15.9 (7.32) | 13.8 (4.81)

6. Primary Outcome: Maximum Observed Concentration (Cmax) of a Single Dose of 5 mg Saxagliptin Versus Cmax of Saxagliptin When Co-administered With 10 mg Dapagliflozin - PK Evaluable Population
Description: Serial blood samples for determination of study drug were collected predose (0 h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Plasma samples were analyzed for saxagliptin by Liquid chromatography-Mass Spectrometry (LC-MS/MS) using a validated method (quantitation range of 0.100 ng/mL to 50.0 ng/mL). Cmax for Saxagliptin was derived from plasma concentration versus time data using a validated PK analysis program ™ and was measured in nanograms per milliliter (ng/mL).
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: PK Evaluable Population: All participants who received at least 1 dose of any study drug and had at least 1 valid PK parameter for at least 1 analyte.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 5 mg Saxagliptin: Treatment A: Single dose Saxagliptin 5mg, Tablet, Oral.
Arm/Group | 5 mg Saxagliptin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 42 | 42
ng/mL | 23.6 (31) | 21.9 (33)
Statistical Analysis 1: Comparison: 5 mg Saxagliptin vs 5 mg Saxagliptin + 10 mg Dapagliflozin; This analysis assesses the effect of concomitant administration of dapagliflozin on the Pharmacokinetics of saxagliptin. The statistical model includes treatment and period as fixed effects and measurements within each participant as repeated measurements. The adjusted geometric means are from the mixed model; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric mean = 0.927, 90% CI 2-sided [0.883 to 0.972]

7. Secondary Outcome: Plasma Apparent Clearance (CLT/F) of a Single Dose of Dapagliflozin Versus CLT/F of Dapagliflozin When Co-administered With Saxagliptin - PK Evaluable Population
Description: Serial blood samples for determination of study drug were collected predose (0 h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Plasma samples were analyzed for dapagliflozin by HPLC-MS/MS using a validated method. Actual sampling times were used for PK calculations. CLT/F was calculated as Dose/AUC(INF)and was measured in milliliters per minute (mL/min).
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | 10 mg Dapagliflozin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 41 | 42
mL/min | 305 (24) | 309 (20)

8. Secondary Outcome: Cmax of 5-Hydroxy (5-OH) Saxagliptin From a Single Dose Saxagliptin Versus Cmax of 5-OH When Saxagliptin Was Co-administered With Dapagliflozin - PK Evaluable Population
Description: Serial blood samples for determination of study drug were collected predose (0 h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Plasma samples were analyzed for 5-OH by LC-MS/MS using a validated method (quantitation range of 0.200 ng/mL to 100.0 ng/mL). Actual sampling times were used for PK calculations. Cmax for 5-OH Saxagliptin (the major active metabolite of Saxagliptin) was derived from plasma concentration versus time data using a validated PK analysis program ™ and was measured in ng/mL.
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 10 mg Dapagliflozin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 42 | 42
ng/mL | 47.0 (30) | 49.6 (27)
Statistical Analysis 1: Comparison: 10 mg Dapagliflozin vs 5 mg Saxagliptin + 10 mg Dapagliflozin; This analysis assesses the effect of concomitant administration of dapagliflozin on the Pharmacokinetics of 5-OH saxagliptin (metabolite of saxagliptin). The statistical model includes treatment and period as fixed effects and measurements within each participant as repeated measurements. The adjusted geometric means are from the mixed model; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric mean = 1.055, 90% CI 2-sided [1.004 to 1.109]

9. Primary Outcome: AUC(0-T) of Saxagliptin From Single Dose 5 mg Saxagliptin Versus AUC(0-T) of Saxagliptin When Co-administered With 10 mg Dapagliflozin - PK Evaluable Population
Description: Serial blood samples for determination of study drug were collected predose (0 h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Plasma samples were analyzed for saxagliptin by Liquid chromatography-Mass Spectrometry (LC-MS/MS) using a validated method (quantitation range of 0.100 ng/mL to 50.0 ng/mL). AUC(0-T), the area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (linear up/log down trapezoidal method) was derived from the plasma concentration versus time profile for study drug using a validated PK analysis program ™ and was measured in nanograms*hours per milliliter (ng*h/mL).
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- 5 mg Saxagliptin: Treatment A: single dose of Saxagliptin 5mg, Tablet, Oral.
Arm/Group | 5 mg Saxagliptin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 42 | 42
ng*h/mL | 87.8 (23) | 87.0 (23)
Statistical Analysis 1: Comparison: 5 mg Saxagliptin vs 5 mg Saxagliptin + 10 mg Dapagliflozin; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric mean = 0.991, 90% CI 2-sided [0.960 to 1.022]

10. Primary Outcome: AUC(INF) of Saxagliptin From a Single Dose of 5 mg Saxagliptin Versus AUC(INF) of Saxagliptin When Co-administered With 10 mg Dapagliflozin - PK Evaluable Population
Description: Serial blood samples for determination of study drug were collected predose (0 h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Plasma samples were analyzed for saxagliptin by LC-MS/MS using a validated method (quantitation range of 0.100 ng/mL to 50.0 ng/mL). AUC(INF) was derived from the plasma concentration versus time profile using a validated PK analysis program ™ and was measured in nanograms*hours per milliliter (ng*h/mL).
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 5 mg Saxagliptin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 42 | 42
ng*h/mL | 89.0 (23) | 88.2 (23)
Statistical Analysis 1: Comparison: 5 mg Saxagliptin vs 5 mg Saxagliptin + 10 mg Dapagliflozin; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric mean = 0.991, 90% CI 2-sided [0.961 to 1.022]

11. Secondary Outcome: AUC(0-T) of 5-OH Saxagliptin From Single Dose Saxagliptin Versus AUC(0-T) of 5-OH From Saxagliptin Co-administered With Dapagliflozin - PK Evaluable Population
Description: Serial blood samples for determination of study drug were collected predose (0 h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Plasma samples were analyzed for 5-OH by LC-MS/MS using a validated method (quantitation range of 0.200 ng/mL to 100.0 ng/mL). AUC(0-T) is area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (linear up/log down trapezoidal method)and was derived from the plasma concentration versus time profile for study drug using a validated PK analysis program ™. AUC (0-T) was measured in nanograms*hours per milliliter (ng*h/mL).
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 10 mg Dapagliflozin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 42 | 42
ng*h/mL | 267 (22) | 289 (22)
Statistical Analysis 1: Comparison: 10 mg Dapagliflozin vs 5 mg Saxagliptin + 10 mg Dapagliflozin; This analysis assesses the effect of concomitant administration of dapagliflozin on the Pharmacokinetics of 5-OH saxagliptin (metabolite). The statistical model includes treatment and period as fixed effects and measurements within each participant as repeated measurements. The adjusted geometric means are from the mixed model; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric mean = 1.085, 90% CI 2-sided [1.058 to 1.113]

12. Secondary Outcome: AUC(INF) of 5-OH Saxagliptin From a Single Dose Saxagliptin Versus AUC(INF) of 5-OH When Saxagliptin Was Co-administered With Dapagliflozin - PK Evaluable Population
Description: Serial blood samples for determination of study drug were collected predose (0 h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Plasma samples were analyzed for 5-OH by LC-MS/MS using a validated method (quantitation range of 0.200 ng/mL to 100.0 ng/mL). AUC(INF) was derived from the plasma concentration versus time profile using a validated PK analysis program ™ and was measured in nanograms*hours per milliliter (ng*h/mL).
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 10 mg Dapagliflozin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 42 | 42
ng*h/mL | 273 (22) | 296 (22)
Statistical Analysis 1: Comparison: 10 mg Dapagliflozin vs 5 mg Saxagliptin + 10 mg Dapagliflozin; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Mixed Models Analysis; ratio of adjusted geometric mean = 1.085, 90% CI 2-sided [1.058 to 1.113]

13. Secondary Outcome: Cmax of the Saxagliptin Total Active Moiety From a Single Dose of 5 mg Saxagliptin Versus Cmax of Saxagliptin Total Active Moiety When Saxagliptin Was Co-administered With 10 mg Dapagliflozin - PK Evaluable Population
Description: Serial blood samples for determination of study drug were collected predose (0 h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Cmax of saxagliptin total active moiety (molar summations of saxagliptin exposure parameter with one-half the molar exposure parameters for 5-OH Saxagliptin) was derived from the plasma concentration versus time profile for the saxagliptin total active moiety. Measurement was in nano Molars (nM).
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Groups:
- 5 mg Saxagliptin: Treatment A: Single dose oral tablet of 5 mg saxagliptin.
Arm/Group | 5 mg Saxagliptin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 42 | 42
nM | 138 (20) | 137 (21)
Statistical Analysis 1: Comparison: 5 mg Saxagliptin vs 5 mg Saxagliptin + 10 mg Dapagliflozin; This analysis assesses the effect of concomitant administration of dapagliflozin on the Pharmacokinetics of saxagliptin total active moiety. The statistical model includes treatment and period as fixed effects and measurements within each participant as repeated measurements. The adjusted geometric means are from the mixed model; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric mean = 0.994, 90% CI 2-sided [0.960 to 1.030]

14. Secondary Outcome: AUC(INF) and AUC(0-T) of the Saxagliptin Total Active Moiety From a Single Dose 5 mg Saxagliptin Versus AUC(INF) and AUC(0-T) of Saxagliptin Total Active Moiety When Saxagliptin Was Co-administered With 10 mg Dapagliflozin - PK Evaluable Population
Description: Serial blood samples for determination of study drug were collected predose (0 h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Plasma samples were analyzed for saxagliptin by LC-MS/MS using a validated method. AUC(INF) is area under the plasma concentration-time curve from time zero extrapolated to infinity; AUC(0-T) is area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (linear up/log down trapezoidal method) and both were derived from the plasma concentration versus time profile using a validated PK analysis program ™. Total moiety (molar summations of saxagliptin exposure parameter with one-half the molar exposure parameters for 5-OH Saxagliptin), AUC(0-T)and AUC(INF) were measured in nano Molars*hours (nM*h).
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM*h
Arm/Group | 5 mg Saxagliptin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 42 | 42
nM*h
  AUC(INF) for Saxagliptin Total Active Moiety | 702 (15) | 735 (15)
  AUC(0-T) for Saxagliptin Total Active Moiety | 694 (15) | 727 (15)
Statistical Analysis 1: Comparison: 5 mg Saxagliptin vs 5 mg Saxagliptin + 10 mg Dapagliflozin; This analysis assesses the effect of concomitant administration of dapagliflozin on the AUC(0-T) of saxagliptin total active moiety. The statistical model includes treatment and period as fixed effects and measurements within each participant as repeated measurements. The adjusted geometric means are from the mixed model; Test type: Superiority or Other; Mixed Models Analysis; Ratio of adjusted geometric mean = 1.046, 90% CI 2-sided [1.029 to 1.064]

15. Secondary Outcome: Tmax of Saxagliptin, 5-OH Saxagliptin, Saxagliptin Total Active Moiety From a Single Dose of Saxagliptin Versus Tmax of Saxagliptin, 5-OH, Saxagliptin Total Active Moiety When Saxagliptin Was Co-administered With Dapagliflozin - PK Evaluable Population
Description: Serial blood samples for determination of study drug were collected predose (0 h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Plasma samples were analyzed for saxagliptin and 5-OH by LC-MS/MS using a validated method. Tmax was derived from the plasma concentration versus time profile for study drug and was measured in hours (h). Saxagliptin was the drug, 5-OH saxagliptin was the metabolite, and Saxagliptin total Active Moiety was molar summations of saxagliptin exposure parameter with one-half the molar exposure parameters for 5-OH Saxagliptin.
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: as for outcome 6
Measure: Median (Full Range); unit: h
Groups:
- 5 mg Saxagliptin: Treatment A: Single saxagliptin 5mg, Tablet, Oral.
Arm/Group | 5 mg Saxagliptin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 42 | 42
h
  Tmax of Saxagliptin | 0.50 [0.50 to 2.00] | 1.00 [0.50 to 2.00]
  Tmax of 5-OH Saxagliptin | 1.50 [1.00 to 2.00] | 1.50 [1.00 to 3.00]
  Tmax of Saxagliptin Total Active Moiety | 1.00 [0.50 to 2.00] | 1.00 [0.50 to 2.00]

16. Secondary Outcome: Half-life (T-HALF) of Saxagliptin, and 5-OH Saxagliptin From Single Dose 5 mg Saxagliptin Versus T-HALF of Saxagliptin and 5-OH From Co-administered Saxagliptin With 10 mg Dapagliflozin - PK Evaluable Population
Description: Serial blood samples for determination of study drug were collected predose (0 h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Plasma samples were analyzed for saxagliptin by LC-MS/MS using a validated method. T-HALF was derived from the plasma concentration versus time profile using a validated PK analysis program ™ and was measured in hours (h).
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 5 mg Saxagliptin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 42 | 42
h
  T-HALF for Saxagliptin | 5.86 (2.23) | 5.38 (2.17)
  T-HALF for 5-OH Saxagliptin | 15.9 (3.06) | 17.0 (2.97)

17. Secondary Outcome: Metabolite to Parent Molar Ratios (MR) of Cmax, AUC(INF), and AUC(0-T) of 5-OH Saxagliptin and Saxagliptin From a Single Dose 5 mg Saxagliptin Versus MR of Saxagliptin and 5-OH When Saxagliptin Was Co-administered With 10 mg Dapagliflozin - PK Evaluable
Description: Serial blood samples for determination of study drug were collected predose (0 h), 6 h, 12 h, 18 h, 24 h, 30 h, 36 h, 42 h, 48 h, 54 h and 60 h postdose, relative to dosing on Day 1 in each cross over period. Saxagliptin is the parent drug and 5-OH saxagliptin is the metabolite. The molecular weights to be used for the molar ratios were 315.42 and 331.42 for saxagliptin and 5-OH, respectively. Plasma samples were analyzed for saxagliptin and for 5-OH by LC-MS/MS using a validated method (quantitation range of 0.100 ng/mL to 50.0 ng/mL and 0.200 ng/mL to 100.0 ng/mL for saxagliptin and 5-OH, respectively).
Time Frame: Day 1 (0h to 60h post dose) in each period
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Molar ratio
Arm/Group | 5 mg Saxagliptin | 5 mg Saxagliptin + 10 mg Dapagliflozin
Number analyzed (Participants) | 42 | 42
Molar ratio
  MR_Cmax | 1.90 (37) | 2.16 (37)
  MR_AUC(INF) | 2.92 (33) | 3.19 (33)
  MR_AUC(0-T) | 2.89 (33) | 3.16 (34)

18. Secondary Outcome: Number of Participants With Deaths, Serious Adverse Events, Adverse Events, or Discontinuations Due to Adverse Events - Safety Population
Description: Adverse event (AE)=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. Serious adverse event (SAE)=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Treatment-related=having certain, probable, possible, or missing relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death. End of study was approximately 16 days and was the time for a participant to conclude each of the 3 periods (including the 6 day washout between periods).
Time Frame: Day 1 to end of study (16 days)
Population: Safety Population = All participants who received at least one dose of any study drug.
Measure: Number; unit: participants
Groups:
- Treatment A: Saxagliptin 5mg: Treatment A: Single dose oral tablet of 5 mg saxagliptin..
- Treatment B: Dapagliflozin 10mg: Treatment B: A single oral tablet dose of 10 mg Dapagliflozin.
- Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg: Treatment C: Co-administration of a single dose oral tablet of 10 mg dapagliflozin plus a single dose of oral tablet of 5mg saxagliptin..
Arm/Group | Treatment A: Saxagliptin 5mg | Treatment B: Dapagliflozin 10mg | Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg
Number analyzed (Participants) | 42 | 42 | 42
participants
  Participants with AEs | 6 | 9 | 8
  Participants with treatment-related AEs | 4 | 4 | 7
  Participants with SAEs | 0 | 0 | 0
  Participants discontinuing due to AEs | 0 | 0 | 0
  Deaths | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Marked Hematology Laboratory Abnormalities - Safety Population
Description: Fasted for 10 hours prior to samples taken. Baseline was Day -1 of Period 1; study drug was administered on Day 1 of each crossover period. Lower limit of normal (LLN); upper limit of normal (ULN); pretreatment(pre-RX); treatment (RX). Hemoglobin (g/L): <0.85* pre-RX; hematocrit (vol): <0.85*pre-RX; erythrocytes (*10^12 c/L): <0.85*pre-RX; platelet count (*10^9 c/L): <0.85*LLN if pre-RX>=LLN, or if Pre-Tx <LLN; leukocytes (*10^9 c/L): <0.85*LLN if pre-RX <LLN,or <0.9*LLN if LLN<=Pre-RX<=ULN; neutrophils+bands (*10^9 c/L): <0.85*Pre-RX if Pre-RX <1.5 or <1.5 if Pre-RX >=1.5; eosinophils (*10^9 c/L): if value >0.75; basophils (*10^9 c/L): if value >0.4; monocytes (*10^9c/L): if value >2; lymphocytes (*10^9 c/L): if value <0.750 or if value >7.50.
Time Frame: Baseline to Day 1 of each period
Population: Safety Population = All participants who received at least one dose of any study drug.
Measure: Number; unit: participants
Groups:
- Treatment A: Saxagliptin 5mg: Single dose oral tablet of 5 mg saxagliptin.
- Treatment B: Dapagliflozin 10mg: A single oral tablet dose of 10 mg Dapagliflozin.
- Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg: Co-administration of a single dose oral tablet of 10 mg dapagliflozin plus a single dose of oral tablet 5mg saxagliptin.
Arm/Group | Treatment A: Saxagliptin 5mg | Treatment B: Dapagliflozin 10mg | Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg
Number analyzed (Participants) | 42 | 42 | 42
participants
  Leukocytes Low | 0 | 0 | 1
  Neutrophils (absolute) Low | 1 | 1 | 1

20. Secondary Outcome: Mean Change From Baseline in Systolic and Diastolic Blood Pressure - Safety Population
Description: Blood pressure was taken while the participant was quietly seated for at least 5 minutes. Blood pressure was measured in millimeters of mercury (mmHg). Baseline was Day -1 in Period 1; study drug was administered on Day 1 of each crossover period.
Time Frame: Baseline to Day 1 of each period
Population: Safety Population = All participants who received at least one dose of any study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Treatment B: Dapagliflozin 10mg: Single dose oral tablet of 10 mg dapagliflozin.
Arm/Group | Treatment A: Saxagliptin 5mg | Treatment B: Dapagliflozin 10mg | Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg
Number analyzed (Participants) | 42 | 42 | 42
mmHg
  Systolic Blood Pressure | -6.0 (7.41) | -4.6 (8.13) | -7.2 (8.35)
  Diastolic Blood Pressure | -2.6 (4.94) | -2.0 (4.86) | -3.3 (6.23)

21. Secondary Outcome: Mean Change From Baseline in Heart Rate - Safety Population
Description: Heart rates were taken while the participant was sitting quietly for at least 5 minutes and were measured in beats per minute (bpm). Baseline was Day -1 of Period 1; study drug was administered on Day 1 of each crossover period.
Time Frame: Baseline to Day 1 in each period
Population: Safety Population = All participants who received at least one dose of any study drug.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Treatment A: Saxagliptin 5mg | Treatment B: Dapagliflozin 10mg | Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg
Number analyzed (Participants) | 42 | 42 | 42
bpm | -4.4 (7.04) | -4.0 (9.64) | -4.3 (10.52)

22. Secondary Outcome: Mean Change From Baseline in Respiration Rate - Safety Population
Description: Respiration rates were taken while the participant was sitting quietly for at least 5 minutes and were measured in breaths per minute (bpm). Baseline was Day -1 of Period 1; study drug was administered on Day 1 of each crossover period.
Time Frame: Baseline to Day 1 in each period
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Treatment A: Saxagliptin 5mg | Treatment B: Dapagliflozin 10mg | Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg
Number analyzed (Participants) | 42 | 42 | 42
bpm | -0.4 (3.46) | -1.2 (2.89) | -0.9 (3.13)

23. Secondary Outcome: Mean Change From Baseline in Temperature - Safety Population
Description: Participant had their temperature taken after quietly sitting for at least 5 minutes and it was measured as degrees of centigrade (C). Baseline was Day -1 of Period 1; study drug was administered on Day 1 of each crossover period.
Time Frame: Baseline to Day 1 in each period
Population: Safety Population = All participants who received at least one dose of any study drug.
Measure: Mean (Standard Deviation); unit: degrees of centigrade
Arm/Group | Treatment A: Saxagliptin 5mg | Treatment B: Dapagliflozin 10mg | Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg
Number analyzed (Participants) | 42 | 42 | 42
degrees of centigrade | -0.15 (0.393) | -0.23 (0.383) | -0.16 (0.385)

24. Secondary Outcome: Number of Participants With Marked Chemistry Laboratory Abnormalities - Safety Population
Description: Fasted for 10 hours prior to samples taken. Baseline was Day -1 of Period 1; study drug was administered on Day 1 of each crossover period. Lower limit of normal(LLN); upper limit of normal (ULN); pre-treatment(Pre-Rx). Alkaline phosphatase U/L:>1.25*Pre-RX if Pre-Rx >ULN or >1.25*ULN if Pre-Rx <=ULN; aspartate aminotransferase (AST) U/L: >1.25*Pre-Rx if Pre-Rx > ULN or 1.25*ULN if Pre-Rx <= ULN;alanine aminotransferase (ALT) U/L: >1.25*Pre-Rx if Pre-Rx>ULN or 1.25*ULN if Pre-Rx<=ULN;blood urea nitrogen (BUN)mmol/L: >1.1*ULN if Pre-Rx <=ULN or >1.2*Pre-Rx if Pre-Rx >ULN; total bilirubin µmol/L: >1.1*ULN if Pre-Rx <=ULN or >1.25*Pre-Rx if Pre-Rx >ULN;direct bilirubin µmol/L: >1.1*ULN if Pre-Rx <= ULN or >1.25*Pre-Rx if Pre-Rx > ULN; creatine phosphokinase (CK) U/L: >1.5*Pre-Rx if Pre-Rx >ULN or >1.5*ULN if Pre-Rx <= ULN.
Time Frame: Baseline to Day 1 in each period
Population: Safety Population = All participants who received at least one dose of any study drug.
Measure: Number; unit: participants
Groups:
- Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg: Co-administration of a single dose oral tablet of 10 mg dapagliflozin plus a single dose of oral tablet of 5mg saxagliptin.
Arm/Group | Treatment A: Saxagliptin 5mg | Treatment B: Dapagliflozin 10mg | Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg
Number analyzed (Participants) | 42 | 42 | 42
participants
  Total Bilirubin High | 1 | 1 | 1
  Direct Bilirubin High | 1 | 1 | 1
  ALT High | 1 | 0 | 1
  BUN High | 1 | 0 | 0
  CK High | 0 | 0 | 1

25. Secondary Outcome: Number of Participants With Marked Urinalysis Laboratory Abnormalities - Safety Population
Description: Baseline was Day -1 of Period 1; study drug was administered on Day 1 of each crossover period. Fasted for 10 hours prior to samples taken. LLN=lower limit of normal; ULN=upper limit of normal; pretreatment (Pre-Rx). Normals: Urine glucose qualitative: dipstick >=1 if Pre-Rx <1 or 2*Pre-Rx if Pre-Rx>=1; urine microscopic white blood cell count (WBC): >=2 if Pre-Rx <2 or >=4 if Pre-Rx >=2;urine red blood cell count (RBC):>=2 if Pre-Rx <2 or >=4 if Pre-Rx >=2.
Time Frame: Baseline to Day 1 of each period
Population: Safety Population = All participants who received at least one dose of any study drug. Urine WBC and RBC were not done for all 42 participants. Number of participants analyzed (N) for the 3 treatments for WBC/RBC urine were 4, 8, 6, in treatment A, B, C, respectively.
Measure: Number; unit: participants
Arm/Group | Treatment A: Saxagliptin 5mg | Treatment B: Dapagliflozin 10mg | Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg
Number analyzed (Participants) | 42 | 42 | 42
participants
  Urine Glucose High (N=42, 42, 42) | 0 | 2 | 5
  Urine WBC and RBC High (N= 4, 8, 6) | 0 | 0 | 1

26. Secondary Outcome: Number of Participants With Change From Baseline in ECG Interval - Safety Population
Description: A 12-Lead electrocardiogram (ECG) was performed and recorded after the participant had been supine for at least 5 minutes. ECGs done at baseline (Day-1 of Period 1) and at end of study; therefore the results are presented by sequence, and cannot be presented by treatment. QT interval (measure between Q wave and T wave in the heart's electrical cycle); and QT interval corrected for heart rate using Fridericia's formula (QTcF) were measured in milliseconds (msec). Abnormality criteria: QT/QTcF QT or QTcF >450 msec and <=480 msec at any postdose time point and not present at baseline. QT or QTcF >480 msec and <=500 msec at any postdose time point and not present at baseline QT or QTcF >500 msec at any postdose time point and not present at baseline. QT/QTcF Increase from baseline >60 msec for at least 1 postdose measurement. Increase from baseline in QT or QTcF >30 msec for at least 1 postdose measurement, but <=60 msec for all postdose measurements.
Time Frame: Baseline to end of study (16 days)
Population: Safety Population = All participants who received at least one dose of any study drug.
Measure: Number; unit: participants
Arm/Group | A-B-C: Saxagliptin-Dapagliflozin-(Saxagliptin+Dapagliflozin) | A-C-B: Saxagliptin-(Saxagliptin+Dapagliflozin)-Dapagliflozin | B-A-C: Dapagliflozin-Saxagliptin-(Saxagliptin+Dapagliflozin) | B-C-A: Dapagliflozin-(Saxagliptin+Dapagliflozin)-Saxagliptin | C-A-B: (Saxagliptin+Dapagliflozin)-Saxagliptin-Dapagliflozin | C-B-A: (Saxagliptin+Dapagliflozin)-Dapagliflozin-Saxagliptin
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7 | 7
participants
  QT change from baseline >60 msec | 0 | 0 | 0 | 1 | 0 | 0
  QT change from baseline >30 msec; <=60 msec | 0 | 4 | 0 | 0 | 0 | 0
  QTcF change from baseline >60 msec | 0 | 0 | 0 | 0 | 0 | 0
  QTcF change from baseline >30 msec; <=60 msec | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day -1 to end of study (approximately 16 days). Total length of 3 crossover periods.
Groups:
- Treatment A: Saxagliptin 5mg: Saxagliptin 5mg, Tablet, Oral, Once daily, 1 day in each of 3 periods.
- Treatment B: Dapagliflozin 10mg: Dapagliflozin 10mg, Tablet, Oral, Once daily, 1 day in each of 3 periods.
- Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg: Saxagliptin 5 mg + Dapagliflozin 10 mg, Tablets, Oral, Once daily, 1 day in each of 3 periods.
Arm/Group | Treatment A: Saxagliptin 5mg | Treatment B: Dapagliflozin 10mg | Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 6/42 | 9/42 | 8/42
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Saxagliptin 5mg (N=42) | Treatment B: Dapagliflozin 10mg (N=42) | Treatment C: Saxagliptin 5 mg + Dapagliflozin 10 mg (N=42)
Headache (Nervous system disorders) | 0 | 2 | 4
Constipation (Gastrointestinal disorders) | 2 | 1 | 2
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0
ALT increased (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.